CLINICAL TRIAL: NCT03937908
Title: A Pharmacokinetic Study of Centella Asiatica Product (CAP) in Elderly Participants With Mild Cognitive Impairment Receiving Cholinesterase Inhibitor Therapy
Brief Title: Pharmacokinetics Centella Asiatica Product (CAP) in Mild Cognitive Impairment
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Participant study visits not possible during COVID-19 pandemic. Funder not able to support a continuation at some future date.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Amala Soumyanath, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00017985; R61AT009628 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-05-06 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Impairment; Elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is an outpatient open-label clinical study using a blinded randomized crossover design of two doses.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will use an arm equivalence design to promote equal numbers of participants for each order schema. All participants will be blinded to the dose they will be receiving at each visit. The investigators have developed a formulation that tastes and looks very similar at each dose. The investigator administering the intervention and the analyst performing the liquid chromatography analysis of collected plasma will be blinded as to the dose of the product administered. The liquid chromatography analyst will also be blinded as to the time point of collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2g CAP (Experimental): Single administration of 2g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
  Interventions: Drug: 2g Centella asiatica water extract product
- 4g CAP (Experimental): Single administration of 4g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
  Interventions: Drug: 4g Centella asiatica water extract product

INTERVENTIONS:
Drug: 2g Centella asiatica water extract product — 2g of Centella asiatica water extract (CAW) in a standardized product containing excipients to improve palatability, color matching and dispersability. The product (CAP) is a powder which will be dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
  Other Names: CAP 2g
  Arms: 2g CAP
Drug: 4g Centella asiatica water extract product — 4g of Centella asiatica water extract (CAW) in a standardized product containing excipients to improve palatability, color matching and dispersability. The product (CAP) is a powder which will be dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
  Other Names: CAP 4g
  Arms: 4g CAP

SUMMARY:
This study will measure the oral bioavailability and pharmacokinetics of known bioactive compounds from a standardized Centella asiatica water extract product (CAP) in mildly demented elders on cholinesterase inhibitor therapy. Compound levels will be measured in human plasma and urine over 10 hours after acute oral administration of two doses of the botanical extract product. The dose giving maximum plasma levels (Cmax)closest to those observed in the investigator's mouse studies, the area under the curve (AUC0-12), as well as the rate of clearance (t ½) of the known compounds and time of maximum concentration (tmax), will be identified. These data will be used to inform decisions on the dosage and dosing frequency for future clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To assess the bioavailability and rate of clearance of Centella asiatica derived compounds in mildly demented elders on cholinesterase inhibitor therapy through a pharmacokinetic study.
2. To determine the acute tolerability of a Centella asiatica product in mildly demented elders on cholinesterase inhibitor therapy.

OUTLINE:

Participants will orally consume a single administration of a standardized Centella asiatica water extract product (CAP). Two doses (2g and 4g CAW) will be administered on separate occasions, at least two weeks apart. The levels of known bioactive compounds present in Centella asiatica will be measured in human plasma and urine over 10 hours after administration of each of the doses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-85, male and female
2. Meet the National Institute of Aging - Alzheimer's Association core clinical criteria for mild cognitive impairment or probable Alzheimer's disease dementia with a Clinical Dementia Rating (CDR) score of 0.5-1 and MMSE score of 20-28
3. Report a history of subjective memory decline with gradual onset and slow progression over the last one year before screening; MUST be corroborated by an informant
4. On cholinesterase inhibitor therapy for Alzheimer's disease (AD) and must be on a stable dose for at least 12 weeks prior to baseline
5. Caregiver/study partner that can accompany participant to all study visits
6. Sufficient English language skills to complete all tests
7. Sufficient vision and hearing to complete all tests
8. No known allergies to Centella asiatica or CAP excipients
9. Willingness to discontinue all botanical dietary supplements for one week prior to and during each study visit
10. Willingness to comply with a 48-hour low plant diet for each study visit
11. Absence of significant depression symptoms (Geriatric Depression Scale-15 score of <12)
12. Body Mass Index (BMI) greater than 17 and less than 35 at screening
13. General health status that will not interfere with the ability to complete the study

Exclusion Criteria:

1. Current smoking, alcohol or substance abuse according to DSM-V criteria
2. Women who are pregnant, planning to become pregnant or breastfeeding
3. Men who are actively trying to conceive a child or planning to within three months of study completion
4. Severe aversion to venipuncture
5. Abnormal laboratory evaluation indicating asymptomatic and untreated urinary tract infection
6. Cancer within the last five years, with the exception of localized prostate cancer (Gleason Grade <3) and non-metastatic skin cancers
7. Comorbid conditions such as diabetes mellitus, kidney failure, liver failure, hepatitis, blood disorders, clinical symptomatic orthostatic hypotension, and unstable or significantly symptomatic cardiovascular disease
8. Significant disease of the central nervous system such as brain tumor, seizure disorder, subdural hematoma, cranial arteritis, or clinically significant stroke
9. Major depression, schizophrenia, or other major psychiatric disorder defined by DSM-V criteria
10. Medications: sedatives (except those used occasionally for sleep), central nervous system active medications that have not been stable for two months (including beta blockers, cimetidine, SSRIs, SNRIs), anticoagulants (i.e. Warfarin), investigational drugs used within five half-lives of baseline visit, systemic corticosteroids, neuroleptics, anti-Parkinsonian agents, narcotic analgesics, nicotine (tobacco, patches, gum, lozenges, etc.), Cannabis sativa (herb or edibles)
11. Non-Alzheimer dementia such as vascular dementia, normal pressure hydrocephalus or Parkinson's disease
12. Mini Mental State Examination (MMSE) score of <20 or >28 or CDR score >1 or zero
13. Unwilling to maintain stable dosage of AD medications throughout study duration
14. Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
15. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amala Soumyanath, PhD, Principal Investigator — OHSU Department of Neurology
Locations (1):
- Oregon Health and Science University Department of Neurology, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
ALL IPD that underlie results in a publication will be shared via a published journal article.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately after publication and for a period of 3 years following publication.
Access Criteria: Anyone who wishes access to the data, for any reason. Requests should be directed to Dr. Amala Soumyanath at soumyana@ohsu.edu

REFERENCES:
- [Background] Wright KM, McFerrin J, Alcazar Magana A, Roberts J, Caruso M, Kretzschmar D, Stevens JF, Maier CS, Quinn JF, Soumyanath A. Developing a Rational, Optimized Product of Centella asiatica for Examination in Clinical Trials: Real World Challenges. Front Nutr. 2022 Jan 14;8:799137. doi: 10.3389/fnut.2021.799137. eCollection 2021. PMID 35096945
- [Result] Wright KM, Bollen M, David J, Speers AB, Brandes MS, Gray NE, Alcazar Magana A, McClure C, Stevens JF, Maier CS, Quinn JF, Soumyanath A. Pharmacokinetics and Pharmacodynamics of Key Components of a Standardized Centella asiatica Product in Cognitively Impaired Older Adults: A Phase 1, Double-Blind, Randomized Clinical Trial. Antioxidants (Basel). 2022 Jan 23;11(2):215. doi: 10.3390/antiox11020215. PMID 35204098

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: 2g CAP Then 4g CAP: Participants first received one single administration of 2g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach. After a washout period of 14 days, they then received one single administration of 4g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
- Experimental: 4g CAP Then 2g CAP: Participants first received one single administration of 4g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach. After a washout period of 14 days, they then received one single administration of 2g of Centella asiatica water extract standardized product dissolved in 10-12 ounce of water and consumed by mouth once on an empty stomach.
Period: Overall Study
Arm/Group | Experimental: 2g CAP Then 4g CAP | Experimental: 4g CAP Then 2g CAP
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Study discontinuation due to pandemic restrictions | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline values for all participants before randomization
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28 (2)
White blood cells [Mean (Standard Deviation); unit: x10^3 cells/uL] | 7.28 (0.60)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 132 (7)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 81 (3)
Body temperature [Mean (Standard Deviation); unit: Celsius] | 36.7 (0.1)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 68 (5)
Red blood cells [Mean (Standard Deviation); unit: x10^6 cells/uL] | 4.64 (0.21)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.3 (0.6)
Hematocrit [Mean (Standard Deviation); unit: percentage] | 44 (2)
Platelets [Mean (Standard Deviation); unit: x10^3 platelets/uL] | 259 (20)
Blood glucose [Mean (Standard Deviation); unit: mg/dL] | 81 (3)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 17 (3)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.1)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.6 (0.1)
Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 26 (3)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 32 (3)
Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 87 (12)
Total protein [Mean (Standard Deviation); unit: g/dL] | 7.7 (0.1)
Albumin [Mean (Standard Deviation); unit: g/dL] | 3.8 (0.1)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 141 (1)
Chloride [Mean (Standard Deviation); unit: mmol/L] | 108 (1)
Total CO^2 [Mean (Standard Deviation); unit: mmol/L] | 29 (1)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 3.8 (0.1)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.3 (0.1)
Anion gap [Mean (Standard Deviation); unit: mEq/L] | 5 (1)

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of Centella Asiatica Bioactive Compounds (Cmax)
Description: Following oral administration of a product made from a water extract of Centella asiatica (CAP), the plasma concentration of Centella asiatica derived bioactive compounds (triterpenes, caffeoylquinic acids, and their metabolites) will be measured in blood samples obtained over a 10 hour period, using high performance liquid chromatography tandem mass spectrometry in order to generate a pharmacokinetic curve, and determine pharmacokinetic parameters (maximum concentration) for each of the two doses (2g and 4g).
Time Frame: A 10-hour post-administration period (15, 30, 45, 60, 90, 120, 150, 180, 240, 360, 480, and 600 minutes).
Population: The pharmacokinetic parameter (Cmax) and time curves was calculated using non-compartmental analysis of plasma concentration versus time data using Excel software PK-solver (version 2.0).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 4 | 4
ng/mL
  Asiatic acid | 124 (29) | 259 (24)
  Caffeic acid | 0.3 (0.2) | 1 (0.1)
  Dihydrocaffeic acid | 1 (0.4) | 2 (0.2)
  Dihydroferulic acid | 11 (5) | 20 (6)
  Dicaffeoylquinic acids | 18 (10) | 3 (0.3)
  Ferulic acid | 1 (0.2) | 1.4 (0.1)
  3-(3-hydroxyphenyl)propionic acid | 32 (18) | 42 (18)
  Isoferulic acid | 0.9 (0.3) | 2 (0.1)
  Madecassic acid | 38 (3) | 63 (10)
  Monocaffeoylquinic acids | 14 (7) | 7 (2)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; Asiatic acid; Test type: Equivalence — Two-sided paired t-tests were used to compare pharmacokinetic and clearance parameters between 2g and 4g doses. A p-value of less than 0.05 was considered statistically significant; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; Caffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.23, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; Dihydrocaffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, t-test, 2 sided — Two-sided paired t-tests were used to compare pharmacokinetic and clearance parameters between 2g and 4g doses. A p-value of less than 0.05 was considered statistically significant
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; Dihydroferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; Ferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.07, t-test, 2 sided
Statistical Analysis 6: Comparison: 2g CAP vs 4g CAP; 3-(3-hydroxyphenyl)propionic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.09, t-test, 2 sided
Statistical Analysis 7: Comparison: 2g CAP vs 4g CAP; Isoferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, t-test, 2 sided
Statistical Analysis 8: Comparison: 2g CAP vs 4g CAP; Madecassic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.10, t-test, 2 sided
Statistical Analysis 9: Comparison: 2g CAP vs 4g CAP; Monocaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.11, t-test, 2 sided

2. Primary Outcome: Time of Maximum Concentration (Tmax)
Description: The time of maximum concentration (Tmax) of the known bioactive compounds and their metabolites will be calculated from the concentrations measured by high performance liquid chromatography tandem mass spectrometry in order to help determine dosage intervals
Time Frame: A 10-hour post-administration period (15, 30, 45, 60, 90, 120, 150, 180, 240, 360, 480 and 600 minutes).
Measure: Mean (Standard Error); unit: hours
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 4 | 4
hours
  Asiatic acid | 2 (0.6) | 2 (0.6)
  Caffeic acid | 4 (2) | 4 (1)
  Dihydrocaffeic acid | 3.25 (0.5) | 3.5 (0.5)
  Dihydroferulic acid | 3.4 (1) | 3.5 (0.5)
  Dicaffeoylquinic acids | 6 (2) | 0.6 (0.3)
  Ferulic acid | 5 (0.6) | 5.5 (0.5)
  3-(3-hydroxyphenyl)propionic acid | 6 (1.4) | 5.5 (1.7)
  Isoferulic acid | 1.3 (0.6) | 1 (0.4)
  Madecassic acid | 2 (0.5) | 2 (0.5)
  Monocaffeoylquinic acids | 4 (2) | 2 (0.4)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; Asiatic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.82, t-test, 2 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; Caffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.40, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; Dihydrocaffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.20, t-test, 2 sided
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; Dihydroferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.48, t-test, 2 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; Ferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.20, t-test, 2 sided
Statistical Analysis 6: Comparison: 2g CAP vs 4g CAP; 3-(3-hydroxyphenyl)propionic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.32, t-test, 2 sided
Statistical Analysis 7: Comparison: 2g CAP vs 4g CAP; Isoferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.35, t-test, 2 sided
Statistical Analysis 8: Comparison: 2g CAP vs 4g CAP; Madecassic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.52, t-test, 2 sided
Statistical Analysis 9: Comparison: 2g CAP vs 4g CAP; Monocaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.13, t-test, 2 sided

3. Primary Outcome: Half-life (t1/2)
Description: The half-life (t1/2) of the known bioactive compounds and their metabolites will be calculated from the plasma concentrations measured by high performance liquid chromatography tandem mass spectrometry to help determine dosage intervals.
Time Frame: A 10-hour post-administration period (15, 30, 45, 60, 90, 120, 150,180, 240, 360, 480, and 600 minutes).
Measure: Mean (Standard Error); unit: hours
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 4 | 4
hours
  Asiatic acid | 3.8 (1) | 2.2 (0.5)
  Caffeic acid | 2.6 (1) | 3.5 (1.2)
  Dihydrocaffeic acid | 4.8 (1.3) | 1.1 (0.4)
  Dihydroferulic acid | 4.5 (1.6) | 2.5 (0.3)
  Dicaffeoylquinic acids | 0 (0) | 3 (2)
  Ferulic acid | 13.4 (5.3) | 7 (1.2)
  3-(3-hydroxyphenyl)propionic acid | 2.3 (0.3) | 1.8 (0.7)
  Isoferulic acid | 8.8 (5.7) | 2.9 (0.6)
  Madecassic acid | 1.7 (0.5) | 1.7 (0.9)
  Monocaffeoylquinic acids | 2 (0.5) | 3 (0.3)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; Asiatic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.34, t-test, 2 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; Dihydrocaffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.08, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; Dihydroferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.23, t-test, 2 sided
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; Ferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.14, t-test, 2 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; 3-(3-hydroxyphenyl)propionic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.28, t-test, 2 sided
Statistical Analysis 6: Comparison: 2g CAP vs 4g CAP; Isoferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.17, t-test, 2 sided
Statistical Analysis 7: Comparison: 2g CAP vs 4g CAP; Madecassic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.98, t-test, 2 sided
Statistical Analysis 8: Comparison: 2g CAP vs 4g CAP; Monocaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.16, t-test, 2 sided

4. Secondary Outcome: Area Under the Curve (AUC) of the Concentration vs Time Profiles of Known Bioactives From Centella Asiatica
Description: Following oral administration of a product made from a water extract of Centella asiatica (CAP), the plasma concentration of Centella asiatica derived bioactive compounds (triterpenes, caffeoylquinic acids, and their metabolites) will be measured in blood samples obtained over a 10 hour period, using high performance liquid chromatography tandem mass spectrometry in order to generate a pharmacokinetic curve, and determine pharmacokinetic parameters (area under the curve) for each of the two doses (2g and 4g).
Time Frame: A 10-hour post-administration period (15, 30, 45, 60, 90, 120, 150,180, 240, 360, 480 and 600 minutes).
Measure: Mean (Standard Error); unit: ng x h/mL
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 4 | 4
ng x h/mL
  Asiatic acid | 364 (114) | 935 (178)
  Caffeic acid | 1 (1) | 3 (0.3)
  Dihydrocaffeic acid | 3 (0.4) | 6 (1)
  Dihydroferulic acid | 42 (18) | 77 (25)
  Dicaffeoylquinic acids | 18 (10) | 6 (4)
  Ferulic acid | 7 (2) | 10 (1)
  3-(3-hydroxyphenyl)propionic acid | 100 (46) | 189 (77)
  Isoferulic acid | 5 (2) | 8 (0.4)
  Madecassic acid | 101 (16) | 187 (48)
  Monocaffeoylquinic acids | 18 (6) | 23 (4)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; Asiatic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.04, t-test, 2 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; Caffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; Dihydrocaffeic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.06, t-test, 2 sided
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; Dihydroferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.08, t-test, 2 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; Dicaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.56, t-test, 2 sided
Statistical Analysis 6: Comparison: 2g CAP vs 4g CAP; Ferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.21, t-test, 2 sided
Statistical Analysis 7: Comparison: 2g CAP vs 4g CAP; 3-(3-hydroxyphenyl)propionic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided
Statistical Analysis 8: Comparison: 2g CAP vs 4g CAP; Isoferulic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided
Statistical Analysis 9: Comparison: 2g CAP vs 4g CAP; Madecassic acid; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.23, t-test, 2 sided
Statistical Analysis 10: Comparison: 2g CAP vs 4g CAP; Monocaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.16, t-test, 2 sided

5. Secondary Outcome: Total Urinary Excretion
Description: All urine produced over the 10 hours post-administration was collected into a single container. The concentration of bioactive compounds from Centella asiatica (triterpenes, caffeoylquinic acids, and their metabolites) was measured in the single total urine sample collected over 10 hours after CAP administration. Urine samples were treated with glucuronidase and sulfatase enzymes to release analyte from conjugated (Phase II metabolite) forms of the analyte. All samples were analyzed using high performance liquid chromatography tandem mass spectrometry. The concentrations obtained were multiplied by total urine volume to obtain the total amount of that analyte excreted. The total amount (free and conjugated forms) in micrograms of of each analyte in the 10h urine sample is reported.
Time Frame: Total 10 hours
Measure: Mean (Standard Error); unit: micrograms
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 4 | 4
micrograms
  Asiatic acid | 3 (4) | 4 (2)
  Dihydrocaffeic acid | 47 (25) | 41 (7)
  Dihydroferulic acid | 145 (60) | 242 (54)
  Ferulic acid | 18 (6) | 24 (5)
  3-(3-hydroxyphenyl)propionic acid | 16 (10) | 13 (7)
  Isoferulic acid | 18 (6) | 24 (5)
  Madecassic acid | 8 (2) | 14 (4)
  Monodicaffeoylquinic acids | 17 (8) | 13 (7)
  Madecassoside | 1 (8) | 7 (3)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; Asiatic acid; Test type: Equivalence — Two-sided paired t-tests were used to compare the ng/mL between the 2g and 4g doses. A p-value of less than 0.05 was considered statistically significant; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; Madecassic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.09, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; Asiaticoside; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.4, t-test, 2 sided
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; Madecassoside; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.6, t-test, 2 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; Monocaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.4, t-test, 2 sided
Statistical Analysis 6: Comparison: 2g CAP vs 4g CAP; Dicaffeoylquinic acids; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.1, t-test, 2 sided
Statistical Analysis 7: Comparison: 2g CAP vs 4g CAP; 3-(3-hydroxyphenyl)propionic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.9, t-test, 2 sided
Statistical Analysis 8: Comparison: 2g CAP vs 4g CAP; Caffeic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.03, t-test, 2 sided
Statistical Analysis 9: Comparison: 2g CAP vs 4g CAP; Ferulic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.9, t-test, 2 sided
Statistical Analysis 10: Comparison: 2g CAP vs 4g CAP; Isoferulic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.6, t-test, 2 sided
Statistical Analysis 11: Comparison: 2g CAP vs 4g CAP; Dihydroferulic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.4, t-test, 2 sided
Statistical Analysis 12: Comparison: 2g CAP vs 4g CAP; Dihydrocaffeic acid; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.8, t-test, 2 sided

6. Secondary Outcome: NRF2 Expression
Description: NRF2 gene expression was measured in peripheral blood mononuclear cells following consumption of 2g and 4g of Centella asiatica water extract product (CAP).
Time Frame: 0, 1, 2, 3, 4, and 6h following study intervention
Measure: Mean (Standard Error); unit: fold change in expression from time 0h
Arm/Group | 2g CAP | 4g CAP
Number analyzed (Participants) | 2 | 2
fold change in expression from time 0h
  0 h | 1 (0) | 1 (0)
  1 h | 2 (0.2) | 2 (0.3)
  2 h | 32 (4) | 5 (2)
  3 h | 22 (9) | 3 (1)
  4 h | 12 (7) | 2 (1)
  6 h | 4 (2) | 1 (0.3)
Statistical Analysis 1: Comparison: 2g CAP vs 4g CAP; 1 hour; Test type: Equivalence — Two-sided paired t-tests were used to compare fold induction between 2g and 4g doses. A p-value of less than 0.05 was considered statistically significant; p = 0.1, t-test, 1 sided
Statistical Analysis 2: Comparison: 2g CAP vs 4g CAP; 2 hours; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.1, t-test, 1 sided
Statistical Analysis 3: Comparison: 2g CAP vs 4g CAP; 3 hours; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.3, t-test, 1 sided
Statistical Analysis 4: Comparison: 2g CAP vs 4g CAP; 4 hours; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.5, t-test, 1 sided
Statistical Analysis 5: Comparison: 2g CAP vs 4g CAP; 6 hours; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.5, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during each study visit, 24 hours following study drug administration at each study visit, and 7 days after study visit two (end of study).
Description: Vital signs, EKG and CMP were monitored at baseline and during the visit. Adverse events were collected using a multi-system adverse events questionnaire during and after the visit.
Arm/Group | 2g CAP | 4g CAP
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2g CAP (N=4) | 4g CAP (N=4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Drowsiness (Psychiatric disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Inability to sit still (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rigidity of any body part (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergy symptoms (Immune system disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Heart racing or irregular beating (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension/elevated blood pressure (Cardiac disorders) | 1 (1) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased urination (Renal and urinary disorders) | 0 (0) | 2 (2)
Sunburn or sensitivity of skin to light (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Generalized pain (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was discontinued before the target number of participants were enrolled due to pandemic-related restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03937908/Prot_SAP_000.pdf